CLINICAL TRIAL: NCT05654285
Title: Enteroendocrine, Pancreatic, and Adipocyte Hormonal Response After the Ingestion of Cola Beverages With Sucrose and Non-nutritive Sweeteners in Healthy Adults. Crossover Randomized Controlled Trial
Brief Title: Enteroendocrine Hormonal Response After the Ingestion of Cola Beverages With Sucrose and Non-nutritive Sweeteners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Cesar Galicia Ayala, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HIM/2016/015 SSA 1221
Record Dates: First submitted 2022-11-25; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Aspartame; acetosulfame; Sucrose; stevioside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple masking was applied, as described below. Participants: The drinks were offered in standardized disposable cups so that the participants could not visually identify the test drink. All beverages were offered at approximately 4°C and participants were asked to consume them within 10 minutes.
  Investigator: All participants received the mineral water (control) in the first study session. Allocation to the remaining 3 interventions was randomized for each participant, and members of the research team who administered the beverages, performed blood sampling, processed samples in the laboratory, or followed participants during the study sessions were unaware of the allocation, that is, the type of drink that was administered to each participant.
  Outcomes Assessor: The investigator who performed the statistical analysis did not have access to the identity of the participants or the allocation of interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Carbonated water (Placebo Comparator): 355ml of an orally ingested carbonated water
  Interventions: Other: Cola beverage with aspartame and acesulfame K; Other: Cola beverage with sucrose and stevia
- Cola beverage with aspartame and acesulfame K (Experimental): 355ml of an orally ingested carbonated cola drink, sweetened with 142mg of aspartame and acesulfame k, combined (soft drink in its commercial presentation)
  Interventions: Other: Cola beverage with aspartame and acesulfame K; Other: Cola beverage with sucrose and stevia
- Cola beverage with sucrose and stevia (Experimental): 355ml of an orally ingested carbonated cola drink, sweetened with 16g of sucrose and 15.62mg of stevia (soft drink in its commercial presentation)
  Interventions: Other: Cola beverage with aspartame and acesulfame K; Other: Cola beverage with sucrose and stevia
- Cola beverage with sucrose (Active Comparator): 355ml of an orally ingested carbonated cola drink, sweetened with 37g of sucrose
  Interventions: Other: Cola beverage with aspartame and acesulfame K; Other: Cola beverage with sucrose and stevia

INTERVENTIONS:
Other: Cola beverage with aspartame and acesulfame K — Before starting the study: Subjects were asked to avoid non-nutritive sweetener consumption for 48 hours prior to the study sessions. A standardized menu of 346 Kcal was prescribed for dinner and fasting for at least 8 hours prior to each study session. A 7-day washout period was left between each study session.
  Session 1: Weight, height, and waist circumference were measured, the BMI was calculated, and sociodemographic data of the participants and information on the habitual consumption of soft drinks were collected.
  In each session: The beverages were offered at approximately 4°C, in standardized disposable cups, and the participants were asked to drink them in a maximum time of 10 minutes. Heart rate, respiratory rate, and blood pressure were measured before the intervention and every 30 minutes during the observation period. The subjects who manifested adverse sensations were referred to receive medical attention and withdrawn from the session.
Other: Cola beverage with sucrose and stevia

SUMMARY:
Introduction: The consumption of non-nutritive sweeteners (NNS) has been increasing in recent years, as an alternative to replace sugars and reduce the additional intake of carbohydrates, with the idea of reducing the risk of developing obesity, metabolic syndrome, and diabetes. However, recent evidence shows that their chronic intake induces endocrine alterations that may have an important contribution to the increase in body weight. Few studies have explored the acute effects of NNS beverage consumption on endocrine response, and to date, the evidence has been inconsistent regarding post-drinking effects and potential health risks.

Objective: To evaluate the effect of 3 different types of cola beverages, compared with carbonated water, on glucose, insulin, glucagon, and appetite-regulating hormones during the first 120 minutes after ingestion.

Methods: A triple-blind, randomized crossover controlled trial was carried out in which 20 healthy adult individuals (10 men and 10 women) were included. With a washout period of one week (7 days) and fasting for 8 hours, each participant consumed orally 355 mL of carbonated water (CAR), and the 3 different cola beverages sweetened with sucrose (SUC), aspartame/acesulfame K (ASP), and sucrose/stevia (STE), in its commercial presentation. The serum levels of glucose, insulin, glucagon, GLP-1, GIP, PYY, leptin, pancreatic polypeptide, and ghrelin were determined during the administration of each one of the drinks before the intake of the drink and later at 30, 60, 90, and 120 minutes.

Statistical analysis: A descriptive analysis of the variables was performed. The global response of glucose, insulin and appetite-regulating hormones was estimated and the Area Under the Curve (AUC) was obtained using a trapezoidal model and analyzed for each outcome by one-factor ANOVA. An ANOVA for repeated measures was performed considering treatment and time as factors, and comparisons were made with the carbonated water as a control using the Bonferroni test. P values less than 0.05 were considered statistically significant.

Ethical considerations: Our institution's Research, Bioethics, and Biosafety committees authorized the project. All the participants were informed about the objective, the procedures, and the possible adverse effects considered within the study, and they signed the informed consent before the start of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation expressed through the signing of informed consent

Exclusion Criteria:

* Pregnancy (date of last menstruation >28 days)
* History of diabetes mellitus or glucose intolerance, endocrinopathies, or pancreatic diseases
* Treatment with medications or supplements that modify glucose and insulin (eg antihypertensives, corticosteroids, hypoglycemic agents, hormonal agents, etc.)
* Gastrointestinal diseases or conditions that alter gastric emptying and intestinal transit
* Hypersensitivity to the compounds that will be used in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

PRIMARY OUTCOMES:
Glucose, insulin, glucagon, glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY), glucose-dependent insulinotropic polypeptide (GIP), pancreatic polypeptide (PP), leptin, and ghrelin | Measurements were made at 0 minute (before the intake of the drink)
  4-5mL of venous blood was obtained from each participant and immediately transferred to the laboratory for analysis. The glucose oxidase technique was implemented to determine serum glucose levels. This technique has high intra- and inter-assay precision (CV: 2.1 and 1.73%, respectively), and high correlation with Gernon's reagent (r=0.993).
  For the determination of insulin, glucagon, GLP-1, PYY, GIP, PP, leptin, and ghrelin levels, implemented the Milliplex Map® immunological assay, which has an intra-assay coefficient of variation of less than 10% and an inter-assay coefficient of less than 15%, with an accuracy greater than 97%.
  The tests were carried out in duplicate.
Glucose, insulin, glucagon, glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY), glucose-dependent insulinotropic polypeptide (GIP), pancreatic polypeptide (PP), leptin, and ghrelin | Measurements were made at 30 minutes after the intake of the drink
  4-5mL of venous blood was obtained from each participant and immediately transferred to the laboratory for analysis. The glucose oxidase technique was implemented to determine serum glucose levels. This technique has high intra- and inter-assay precision (CV: 2.1 and 1.73%, respectively), and high correlation with Gernon's reagent (r=0.993).
  For the determination of insulin, glucagon, GLP-1, PYY, GIP, PP, leptin, and ghrelin levels, implemented the Milliplex Map® immunological assay, which has an intra-assay coefficient of variation of less than 10% and an inter-assay coefficient of less than 15%, with an accuracy greater than 97%.
  The tests were carried out in duplicate.
Glucose, insulin, glucagon, glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY), glucose-dependent insulinotropic polypeptide (GIP), pancreatic polypeptide (PP), leptin, and ghrelin | Measurements were made at 60 minutes after the intake of the drink
  4-5mL of venous blood was obtained from each participant and immediately transferred to the laboratory for analysis. The glucose oxidase technique was implemented to determine serum glucose levels. This technique has high intra- and inter-assay precision (CV: 2.1 and 1.73%, respectively), and high correlation with Gernon's reagent (r=0.993).
  For the determination of insulin, glucagon, GLP-1, PYY, GIP, PP, leptin, and ghrelin levels, implemented the Milliplex Map® immunological assay, which has an intra-assay coefficient of variation of less than 10% and an inter-assay coefficient of less than 15%, with an accuracy greater than 97%.
  The tests were carried out in duplicate.
Glucose, insulin, glucagon, glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY), glucose-dependent insulinotropic polypeptide (GIP), pancreatic polypeptide (PP), leptin, and ghrelin | Measurements were made at 90 minutes after the intake of the drink
  4-5mL of venous blood was obtained from each participant and immediately transferred to the laboratory for analysis. The glucose oxidase technique was implemented to determine serum glucose levels. This technique has high intra- and inter-assay precision (CV: 2.1 and 1.73%, respectively), and high correlation with Gernon's reagent (r=0.993).
  For the determination of insulin, glucagon, GLP-1, PYY, GIP, PP, leptin, and ghrelin levels, implemented the Milliplex Map® immunological assay, which has an intra-assay coefficient of variation of less than 10% and an inter-assay coefficient of less than 15%, with an accuracy greater than 97%.
  The tests were carried out in duplicate.
Glucose, insulin, glucagon, glucagon-like peptide-1 (GLP-1), peptide tyrosine tyrosine (PYY), glucose-dependent insulinotropic polypeptide (GIP), pancreatic polypeptide (PP), leptin, and ghrelin | Measurements were made at 120 minutes after the intake of the drink
  4-5mL of venous blood was obtained from each participant and immediately transferred to the laboratory for analysis. The glucose oxidase technique was implemented to determine serum glucose levels. This technique has high intra- and inter-assay precision (CV: 2.1 and 1.73%, respectively), and high correlation with Gernon's reagent (r=0.993).
  For the determination of insulin, glucagon, GLP-1, PYY, GIP, PP, leptin, and ghrelin levels, implemented the Milliplex Map® immunological assay, which has an intra-assay coefficient of variation of less than 10% and an inter-assay coefficient of less than 15%, with an accuracy greater than 97%.
  The tests were carried out in duplicate.

CONTACTS AND LOCATIONS:
Overall Officials: America L Miranda-Lora, PhD, Study Director — Epidemiological research unit of Endocrinology and nutrition, HIMFG; Miguel Klünder-Klünder, PhD, Study Chair — Deputy director of research management, HIMFG; Cesar Galicia-Ayala, Master, Principal Investigator — Nursing research unit, HIMFG; Armando Vilchis-Ordoñez, PhD, Study Chair — Clinical lab, HIMFG; Briceida López-Martínez, PhD, Study Chair — Clinical lab, HIMFG

IPD SHARING:
Plan to Share IPD: No